CLINICAL TRIAL: NCT04316962
Title: Cancer Rehabilitation in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Norwegian Extra Foundation for Health and Rehabilitation (Other); Askøy Municipality (Unknown)
Responsible Party: Principal Investigator, May Aasebø Hauken, Professor, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: F322
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Cancer Survivors; All Cancers
Keywords: Cancer survivors; Complex rehabilitation; Mixed method; Adults; Longitudinal; Pilot; Feasibility; Adherence; Quality of life; Participation

STUDY DESIGN:
Intervention Model Description: A pilot study using mixed method with a longitudinal explanatory pre-post design, whereby quantitative data are collected longitudinal and qualitative data are collected in means of focus groups at the end of the rehabilitation program (after 12 weeks). Mixed methods design are reckoned to be a new and important research paradigm because the use of both quantitative and qualitative data may provide an increased insight in both processes and outcomes and thereby provide a more nuanced and complete understanding of the topic in focus, here, cancer rehabilitation.
Masking Description: No masking: only single group pre-post
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complex rehabilitation (Experimental): See intervention described elsewhere.
  Interventions: Other: Complex cancer rehabilitation

INTERVENTIONS:
Other: Complex cancer rehabilitation — The program is conducted as group rehabilitation, organized by four hour weekly over 12 weeks (approximately 50 hours) with 8-10 participants in each group over three years. The program is located in Askøy Municipality's 'Health Central' and conducted by a multidisciplinary team.
  The content of the program is based on prior research and clinical experience, consisting of five elements:
  1. Individual goal-setting
  2. Physical activity (2 hours/week) focusing on balance/coordination, cardio and strength.
  3. Psychoeducation: Five teaching sessions and discussions focusing on physical activity, fatigue and late-effects, nutrition, coping, social support and work/studies. In addition, two sessions (first and last) will also include next of kin.
  4. Individual follow-up: Mandatory session at the start and end of the program, otherwise based on individual request and need.
  5. Peer support.

SUMMARY:
More than 70 % of Norwegian cancer patients become longtime survivors. Even if research documents that a large number strive with physical and psychosocial late effects from cancer and cancer treatment, cancer rehabilitation is not an integrated part of the cancer trajectory. Especially, there is a lack of knowledge and research based cancer rehabilitation in primary health care. In this study, the researchers pilot a cancer rehabilitation program in primary health care using a mixed method with a longitudinal pre-post design and focus group interviews. The overall goal is to study the program's feasibility and adherence, as well as outcomes on quality of life and participation. The project will provide new and important knowledge of cancer rehabilitation in primary health care, as well as important knowledge in on planning and designing a larger RCT study on the topic.

DETAILED DESCRIPTION:
This study focuses on piloting a cancer rehabilitation program for cancer survivors (18-70 years of age), conducted in primary health care in a Norwegian municipality. In Norway, more than 70 % of all cancer patients will be long time survivors. However, research documents that cancer survivors are at increased risk for physical and psychosocial late effects with negative consequences for survival, long-time health and quality of life. Still, there is a huge gap between cancer survivors' documented late-effects and unmet needs and cancer rehabilitation interventions.

Background

Current cancer treatment is usually multimodal, hard and long-lasting, whereby many cancer patients experience physical and psychosocial late-effects and challenges. Some late-effects are life threatening, such as cancer relapse, new cancers, or development of chronical diseases. Other late effects influence the individual's health and quality of life negatively, as for example pain, lymphedema, gastrointestinal problems, memory, concentration and cognitive problems, neuropathies, anxiety and depression etc. In addition, cancer survivors report of social, economic and work related challenges. However, fatigue is the most distressing late-effect reported by cancer survivors, as it influences all areas of life, and is regarded as a strong and independent predictor for impaired quality of life.

Even if Norwegians' right to rehabilitation is assigned by law and cancer rehabilitation is a national focus area, cancer rehabilitation is not an integrated part of the cancer trajectory. Research indicate that healthcare providers have limited knowledge of cancer survivors' multidimensional challenges and effective elements in cancer rehabilitation. Consequently, cancer survivors experience lack of information about late-effects, inadequate follow-up and lack of understanding related to their physical and psychosocial challenges, as well as multidimensional rehabilitation interventions. Based on the law, cancer rehabilitation preferably should be conducted in municipalities nearby the patient's home. However, the few existing programs are criticized for being random, fragmented, not research based, only including single elements, and that survivors have to find such offers for themselves. This highlights the need to developed and pilot evidence based cancer rehabilitation programs - especially in primary health care.

Cancer rehabilitation is defined as processes that support cancer survivors to achieve maximal physical, psychological, social and work function within the frames created by cancer and cancer treatment. Consequently, cancer rehabilitation builds on a bio-psychosocial view of health and health promotion.

Even if cancer rehabilitation is a relatively new research field, research shows that effective elements in cancer rehabilitation are based on physical activity and psychosocial interventions. Physical activity is the single element with most evidence, showing positive effects on physical fitness, general health, quality of life, fatigue and return to work for most cancers and ages. Guidelines for cancer survivors recommend moderate physical activity 30 minutes a day, five days a week or more - and physical exercise as a combination of cardiovascular and strength exercise with gradual increase. Different types of psychosocial education have also shown effect on coping and stress reduction in cancer survivors. Such interventions, often called psychoeducation, most often include several elements such as education and illness specific information, emotional support, coping strategies, relaxing technics and discussions. Because cancer survivors challenges are multidimensional and individual, meeting the individual's need are crucial. Consequently, individual follow-up and goal setting are important means in promoting motivation, control and coping expectations that may promote positive physical and psychosocial health.Furthermore, research documents the importance of peer support in cancer rehabilitation, whereby peer support may promote positive changes, psychosocial function, empowerment and quality of life. New research indicates that a multidimensional approach in cancer rehabilitation that combines physical and psychosocial elements are more effective than single interventions related to physical function, quality of life, fatigue and distress. Research also indicate that positive effects of complex interventions are related to group rehabilitation after primary cancer treatment is finished, programs lasting more than three weeks, including several diagnosis and a multidisciplinary approach. Even if most of this research is conducted as in-rehabilitation in the specialist health care level, it seems evident that a complex rehabilitation program in primary healthcare should combine elements of physical activity, psychoeducation, peer support, goal setting and individual follow up for cancer survivors with different types of cancers after completion of primary cancer treatment.

Study goal and research questions

The overall goal of this pilot study is to increase the understanding and knowledge of cancer rehabilitation in primary health care by pilot testing a complex cancer rehabilitation program. Based on this, we have the following research questions:

1. What characterize the psychosocial health and what is participants motivation to attend the program?
2. How are the program's feasibility and adherence?
3. In what degree do the participants achieve their goals and do this lead to increased participation?
4. What are the participants' outcome on physical fitness?
5. What are the participants' short (12 weeks) and long-term outcomes (6 and 12 months) related to quality of life, physical function, fatigue and mental health?
6. What are the participants' experience of the rehabilitation process and what are the participants' recommendations for future programs?

ELIGIBILITY:
Inclusion Criteria:

1. Cancer survivors with any type of cancer
2. Aged 18- 70 years
3. Finished primary cancer treatment within the last three months to five years 4) referred to the study by oncologist or general practitioner assuring the need for, and capability to, to participate in the program

5) Able to speak and read Norwegian

Exclusion Criteria:

1. Severe physical and/or mental comorbidity representing a contraindication for rehabilitation
2. Insufficient cognitive or Language skills to answer study questionnaires and perform interviews.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life after cancer rehabilitation | Change from baseline (T1) to the end of the program = 12 weeks after baseline (T3)
  Self reported quality of life scale: European Organization for Research and Treatment of Cancer (EORTC QLQ C30), 30 questions, 4-point Likert scale 0-3 for 28 items, 0-6 for two items, total score 0-100 (100=highest Level of function/best score)
Participation | Change from baseline (T1) to the end of the program=12 weeks after baseline (T3)
  Participation scale (goal achievement) administrated by professionals: Canadian Occupational Performance Measure (COPM): Participants rate problems in the three areas of self-care, productivity and leisure. Then they rate the importance of each problem and score performance and satisfaction with performance on a 10-point scale ranging from 1 ('not able to do it' or 'not satisfied at all') to 10 ('able to do it extremely well' or 'extremely satisfied').

SECONDARY OUTCOMES:
Long term change in Quality of life | Change from baseline (T1) to 58 weeks (T8= 1 year after end of cancer rehabilitation)
  Self reported quality of life scale: European Organization for Research and Treatment of Cancer (EORTC QLQ C30), 30 questions, 4-point Likert scale 0-3 for 28 items, 0-6 for two items, total score 0-100 (100=highest Level of function/best score)
Physical fitness | Change masured in meters from baseline (T1) to the end of program=12 weeks after baseline (T3)
  6 minutes walking test: Participant walk a predefined route, walk for 6 minutes and number of meter are measured.
Fatigue | Short and longtime change from baseline (T1) to end of program= 12 weeks after baseline (T3); and to six months and one year after end of program (T4 and T5)
  Self reported fatigue scale: Fatigue Questionnaire (FQ), 13 items, whereby 7 items measure physical fatigue, 4 items measure mental fatigue, and two items are related to timeframe. 4-point Likert scale for all items scored from 0-4. Sum score > 4 and more than 6 months duration are defined as fatigue.
Mental Health | Short and longtime change from baseline (T1) to the end of program = 12 weeks after baseline (T3); and to six months and one year after program (T4 and T5)
  Self reported mental health scale: Hospital Anxiety and Depression Scale (HADS), including 7 questions of anxiety (HADS -A) and seven question of depression (HADS-B). Scored on a 4-point Likert Scale (0-4) where a sum score of 11 or more are defined as anxiety/depression.
Work and leisure | Short and longtime change from baseline (T1) to the end of program = 12 weeks after baseline (T3); and to six months and one year after program (T4 and T5)
  Self-reported work/leisure scale: Work and Social Adjustment Scale (WSAS) with five questions, 8- point Likert Scale from 0 (not impaired at all) to 8 (seriously impaired). Max sum score = 40 (seriously impaired function), where scores > 20 indicates seriously psychopathology and scores 10- 20 is associated with significant impaired function.
Feasibility/adherence | Through study completion, on average of 1 year
  Registration of study flow during the program: attendance on physical exercise, physical testing, attendance of psychoeducation sessions, dropout (number/reason), adverse events and missing data in questionaires

OTHER OUTCOMES:
Satisfaction with program | At the end of the program = 12 weeks after baseline (T3)
  Self-reported satisfaction with program: 7 questions, measured on a 4-point Likert scale measuring satisfaction with the content and structure of the program ranging from 0 (not satisfied at all) to 3 (Very satisfied)
Patients' experiences | At the end of the program = 12 weeks after baseline (T3)
  Focus group interviews with a semi-structured interview guide focusing on motivation for the program, satisfaction with content and structure, importance and experienced outcome.
Posttraumatic Growth | Short and longtime change from baseline (T1) to the end of program= 12 weeks after baseline (T3); and to six months and one year after program (T4 and T5)
  Self-reported scale on posttraumatic growth: The Posttraumatic Growth Inventory Short Form (PTGI-SF) with 10 questions measured on a 6-point Likert scale ranging from 0 (not experienced) to 5 (to a very large extent). Max sum score = 50 where higher score indicate higher personal growth.

CONTACTS AND LOCATIONS:
Overall Officials: May Aa Hauken, Professor, Principal Investigator — Center for Crisis Psychology, University of Bergen
Locations (2):
- Norway (2):
  - Center for Crisis Psychology, University of Bergen, Bergen, Vestland
  - Askøy Municipality, Bergen, Vestland

IPD SHARING:
Plan to Share IPD: Yes
We plan to make IPD available to other researchers on NSD (Norwegian Scientific Data)
Supporting Information: Study Protocol, ICF
Time Frame: After the study has finished, earliest in December 2024
Access Criteria: On request

REFERENCES:
- [Background] Cancer Registry of Norway. Cancer in Norway 2018 - Cancer incidence, mortality, survival and prevalence in Norway. Oslo: Cancer Registry of Norway; 2019.
- [Background] Bennion AE, Molassiotis A. Qualitative research into the symptom experiences of adult cancer patients after treatments: a systematic review and meta-synthesis. Support Care Cancer. 2013 Jan;21(1):9-25. doi: 10.1007/s00520-012-1573-x. Epub 2012 Sep 13. PMID 22972487
- [Background] Bibby H, White V, Thompson K, Anazodo A. What Are the Unmet Needs and Care Experiences of Adolescents and Young Adults with Cancer? A Systematic Review. J Adolesc Young Adult Oncol. 2017 Mar;6(1):6-30. doi: 10.1089/jayao.2016.0012. Epub 2016 Jul 25. PMID 27454408
- [Background] Stricker CT, Jacobs LA. Physical late effects in adult cancer survivors. Oncology (Williston Park). 2008 Jul;22(8 Suppl Nurse Ed):33-41. PMID 19856569
- [Background] Brearley SG, Stamataki Z, Addington-Hall J, Foster C, Hodges L, Jarrett N, Richardson A, Scott I, Sharpe M, Stark D, Siller C, Ziegler L, Amir Z. The physical and practical problems experienced by cancer survivors: a rapid review and synthesis of the literature. Eur J Oncol Nurs. 2011 Jul;15(3):204-12. doi: 10.1016/j.ejon.2011.02.005. Epub 2011 Apr 13. PMID 21489873
- [Background] Hewitt M, Greenfield S, Stovall Ee. From cancer patient to cancer survivor. Lost in transition: Institute of Medicine and National Research Council; 2006.
- [Background] Hellbom M, Bergelt C, Bergenmar M, Gijsen B, Loge JH, Rautalahti M, Smaradottir A, Johansen C. Cancer rehabilitation: A Nordic and European perspective. Acta Oncol. 2011 Feb;50(2):179-86. doi: 10.3109/0284186X.2010.533194. PMID 21231779
- [Background] Harrington CB, Hansen JA, Moskowitz M, Todd BL, Feuerstein M. It's not over when it's over: long-term symptoms in cancer survivors--a systematic review. Int J Psychiatry Med. 2010;40(2):163-81. doi: 10.2190/PM.40.2.c. PMID 20848873
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Ewertz M, Jensen AB. Late effects of breast cancer treatment and potentials for rehabilitation. Acta Oncol. 2011 Feb;50(2):187-93. doi: 10.3109/0284186X.2010.533190. PMID 21231780
- [Background] Soon J, Anton A, Torres J, et al. The Spectrum of Late Effects in Survivors of Stage I Seminoma: A Systematic Review. Asia-Pacific Journal of Clinical Oncology. Aug 2017;13:73-73.
- [Background] Bifulco G, De Rosa N, Tornesello ML, Piccoli R, Bertrando A, Lavitola G, Morra I, Di Spiezio Sardo A, Buonaguro FM, Nappi C. Quality of life, lifestyle behavior and employment experience: a comparison between young and midlife survivors of gynecology early stage cancers. Gynecol Oncol. 2012 Mar;124(3):444-51. doi: 10.1016/j.ygyno.2011.11.033. Epub 2011 Nov 23. PMID 22119994
- [Background] Bilodeau K, Tremblay D, Durand MJ. Exploration of return-to-work interventions for breast cancer patients: a scoping review. Support Care Cancer. 2017 Jun;25(6):1993-2007. doi: 10.1007/s00520-016-3526-2. Epub 2017 Jan 4. PMID 28054145
- [Background] Bevilacqua LA, Dulak D, Schofield E, Starr TD, Nelson CJ, Roth AJ, Holland JC, Alici Y. Prevalence and predictors of depression, pain, and fatigue in older- versus younger-adult cancer survivors. Psychooncology. 2018 Mar;27(3):900-907. doi: 10.1002/pon.4605. Epub 2018 Jan 25. PMID 29239060
- [Background] Campos MPO, Hassan BJ, Riechelmann R, Del Giglio A. Cancer-related fatigue: a practical review. Ann Oncol. 2011 Jun;22(6):1273-1279. doi: 10.1093/annonc/mdq458. Epub 2011 Feb 16. PMID 21325448
- [Background] Buffart LM, Ros WJ, Chinapaw MJ, Brug J, Knol DL, Korstjens I, van Weert E, Mesters I, van den Borne B, Hoekstra-Weebers JE, May AM. Mediators of physical exercise for improvement in cancer survivors' quality of life. Psychooncology. 2014 Mar;23(3):330-8. doi: 10.1002/pon.3428. Epub 2013 Oct 14. PMID 24123482
- [Background] The Norwegian Department of Health.2018. Living with cancer. National Cancer Strategy 2018-2022. Oslo
- [Background] Silver JK. Integrating Rehabilitation Into the Cancer Care Continuum. PM R. 2017 Sep;9(9 Suppl 2):S291-S296. doi: 10.1016/j.pmrj.2017.07.075. No abstract available. PMID 28942903
- [Background] Hall AE, Boyes AW, Bowman J, Walsh RA, James EL, Girgis A. Young adult cancer survivors' psychosocial well-being: a cross-sectional study assessing quality of life, unmet needs, and health behaviors. Support Care Cancer. 2012 Jun;20(6):1333-41. doi: 10.1007/s00520-011-1221-x. Epub 2011 Jul 1. PMID 21720746
- [Background] Dahl L, Wittrup I, Vaeggemose U, Petersen LK, Blaakaer J. Life after gynecologic cancer--a review of patients quality of life, needs, and preferences in regard to follow-up. Int J Gynecol Cancer. 2013 Feb;23(2):227-34. doi: 10.1097/IGC.0b013e31827f37b0. PMID 23314284
- [Background] Thorsen L, Gjerset GM, Loge JH, Kiserud CE, Skovlund E, Flotten T, Fossa SD. Cancer patients' needs for rehabilitation services. Acta Oncol. 2011 Feb;50(2):212-22. doi: 10.3109/0284186X.2010.531050. PMID 21231783
- [Background] Stout NL, Silver JK, Raj VS, Rowland J, Gerber L, Cheville A, Ness KK, Radomski M, Nitkin R, Stubblefield MD, Morris GS, Acevedo A, Brandon Z, Braveman B, Cunningham S, Gilchrist L, Jones L, Padgett L, Wolf T, Winters-Stone K, Campbell G, Hendricks J, Perkin K, Chan L. Toward a National Initiative in Cancer Rehabilitation: Recommendations From a Subject Matter Expert Group. Arch Phys Med Rehabil. 2016 Nov;97(11):2006-2015. doi: 10.1016/j.apmr.2016.05.002. Epub 2016 May 27. PMID 27237580
- [Background] Brandenbarg D, Korsten JHWM, Berger MY, Berendsen AJ. The effect of physical activity on fatigue among survivors of colorectal cancer: a systematic review and meta-analysis. Support Care Cancer. 2018 Feb;26(2):393-403. doi: 10.1007/s00520-017-3920-4. Epub 2017 Oct 23. PMID 29058127
- [Background] Burke S, Wurz A, Bradshaw A, Saunders S, West MA, Brunet J. Physical Activity and Quality of Life in Cancer Survivors: A Meta-Synthesis of Qualitative Research. Cancers (Basel). 2017 May 20;9(5):53. doi: 10.3390/cancers9050053. PMID 28531109
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Hartmann U, Muche R, Reuss-Borst M. Effects of a step-by-step inpatient rehabilitation programme on quality of life in breast cancer patients. A prospective randomised study. Onkologie. 2007 Apr;30(4):177-82. doi: 10.1159/000099989. Epub 2007 Mar 23. PMID 17396040
- [Background] Faller H, Schuler M, Richard M, Heckl U, Weis J, Kuffner R. Effects of psycho-oncologic interventions on emotional distress and quality of life in adult patients with cancer: systematic review and meta-analysis. J Clin Oncol. 2013 Feb 20;31(6):782-93. doi: 10.1200/JCO.2011.40.8922. Epub 2013 Jan 14. PMID 23319686
- [Background] Fors EA, Bertheussen GF, Thune I, Juvet LK, Elvsaas IK, Oldervoll L, Anker G, Falkmer U, Lundgren S, Leivseth G. Psychosocial interventions as part of breast cancer rehabilitation programs? Results from a systematic review. Psychooncology. 2011 Sep;20(9):909-18. doi: 10.1002/pon.1844. Epub 2010 Sep 6. PMID 20821803
- [Background] Lauver D, Connolly-Nelson K, Vang P. Health-related goals in female cancer survivors after treatment. Cancer Nurs. 2007 Jan-Feb;30(1):9-15. doi: 10.1097/00002820-200701000-00002. PMID 17235214
- [Background] Scott DA, Mills M, Black A, Cantwell M, Campbell A, Cardwell CR, Porter S, Donnelly M. Multidimensional rehabilitation programmes for adult cancer survivors. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD007730. doi: 10.1002/14651858.CD007730.pub2. PMID 23543556
- [Background] Juvet LK, Elvsaas IKO, Leivseth G, Anker G, Bertheussen GF, Falkmer U, Fors EA, Lundgren S, Oldervoll LM, Thune I, Norderhaug IN. Rehabilitation of Breast Cancer Patients [Internet]. Oslo, Norway: Knowledge Centre for the Health Services at The Norwegian Institute of Public Health (NIPH); 2009 Mar. Report from Norwegian Knowledge Centre for the Health Services (NOKC) No. 02-2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK464742/ PMID 29319956
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Spence RR, Heesch KC, Brown WJ. Exercise and cancer rehabilitation: a systematic review. Cancer Treat Rev. 2010 Apr;36(2):185-94. doi: 10.1016/j.ctrv.2009.11.003. Epub 2009 Dec 4. PMID 19962830
- [Background] Hauken MA, Larsen TMB, Holsen I. "Back on Track": A Longitudinal Mixed Methods Study on the Rehabilitation of Young Adult Cancer Survivors. Journal of Mixed Methods Research. 2017;13(3):339-360.
- [Result] Ahmedzai HH, Oldervoll LM, Sweetmore AH, Hauken MA. Community-Based Multidimensional Cancer Rehabilitation in Norway: A Feasibility Study. Cancer Nurs. 2024 Mar-Apr 01;47(2):E123-E133. doi: 10.1097/NCC.0000000000001161. Epub 2022 Dec 11. PMID 36066332
- [Result] Loken OU, Hauken MA. A Qualitative Study of Cancer Survivors' Experienced Outcomes of a Multidimensional Rehabilitation Program in Primary Healthcare. Cancer Nurs. 2022 May-Jun 01;45(3):E646-E654. doi: 10.1097/NCC.0000000000000989. Epub 2021 Sep 3. PMID 34310389